CLINICAL TRIAL: NCT02817230
Title: Effect of Statins on Epigenetic Reprogramming of Monocytes in Patients With Elevated Levels of LDL
Brief Title: Effect of Statins on Trained Immunity
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-1340
Record Dates: First submitted 2016-06-15; First posted 2016-06-29 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-06

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients referred to the out-patient clinic with LDL levels >4.9 mmol/l
  Interventions: Drug: Statin
- Controls: Matched normocholesterolemic control subjects

INTERVENTIONS:
Drug: Statin
  Groups: Patients

SUMMARY:
In this study, the investigators will determine whether patients with elevated levels of LDL are characterized by specific epigenetic changes in circulating cells of the innate immune system, compared to control subjects with healthy levels of LDL and whether regular statin treatment influences these changes.

DETAILED DESCRIPTION:
Rationale: The innate immune system plays a pivotal role in the development and progression of atherosclerosis. Recently, it was reported that monocytes can develop a long-lasting immunological memory after stimulation with various microorganisms, which has been termed 'trained innate immunity'. This memory is induced by epigenetic reprogramming. Here the investigators hypothesize that monocytes of patients with elevated LDL cholesterol levels show epigenetic changes compared to normocholesterolemic subjects and that this can be reversed by treatment with statins.

Objective: The main objective is to study whether patients with elevated levels of LDL show increased Histone 3 Lysine 4 trimethylation in the promoter regions of pro-inflammatory cytokines and have an augmented ex vivo Toll-Like Receptor agonist-induced cytokine production in isolated monocytes compared to controls. Subsequently the investigators will study the effect of treatment with statins on these responses.

Study design: Observational study Study population: Subjects aged >18 years who have been referred to the out-patient clinic and have LDL levels that require lipid lowering treatment and matched normocholesterolemic control subjects.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* 18 years or older
* Elevated LDL levels (>4.9 mmol/l)
* No previous cardiovascular events

Controls:

* Age > 18 years
* LDL cholesterol < 3.5 mmol/l
* No previous cardiovascular events

Exclusion Criteria:

* Current lipid lowering treatment
* Known malignant disorders, auto-immune disorder, or diabetes
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study
* Clinical signs of acute infection
* Use of anti-inflammatory medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged >18 years who have been referred to the out-patient clinic and have LDL levels that require lipid lowering treatment (LDL>4.9 mmol/l)
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in histone methylation levels in circulating monocytes | Baseline-3 months follow up
  Histone methylation levels on different lysines of histone 3 will be analyzed at baseline and after 3 months of statin treatment

SECONDARY OUTCOMES:
Inflammatory phenotype | Baseline-3 months follow up

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Academic Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam